CLINICAL TRIAL: NCT00793975
Title: Phase I Study of Weekly Anti-Vascular Endothelial Growth Factor Receptor 2 (VEGFR-2) Monoclonal Antibody IMC-1121B in Patients With Advanced Solid Tumors Who Have Not Responded to Standard Therapy
Brief Title: Study of IMC-1121B in Patients With Tumors That Have Not Responded to Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 13918; CP12-0401 (Other: ImClone Systems); I4T-IE-JVBM (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-11-14; First posted 2008-11-19 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Advanced Solid Tumors
Keywords: Tumors; Antibodies, Monoclonal
MeSH Terms: conditions — Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-1121B (Experimental): All patients will receive intravenous infusions of IMC-1121B with the dose depending on which cohort they are enrolled into. A minimum of three patients will be enrolled in each cohort.
  A completed patient will be either a patient who completes the 4-week treatment cycle and 2-week observation period (for a total of 6 weeks), or a patient who discontinues therapy for an IMC-1121B-related toxicity. Toxicity data for each cohort will be reviewed prior to dose escalation.
  When all patients complete a cohort, dose escalation to the next cohort will occur.
  Interventions: Biological: IMC-1121B; Biological: 1121B

INTERVENTIONS:
Biological: IMC-1121B — Cohort 1
  2 mg/kg I.V. once a week for 4 weeks, followed by a 2-week observation period.
Biological: 1121B — Cohort 2
  4 mg/kg I.V. once a week for 4 weeks, followed by a 2-week observation period.
Biological: 1121B — Cohort 3
  6 mg/kg I.V. once a week for 4 weeks, followed by a 2-week observation period.
Biological: 1121B — Cohort 4
  8 mg/kg I.V. once a week for 4 weeks, followed by a 2-week observation period.
Biological: 1121B — Cohort 5
  10 mg/kg I.V. once a week for 4 weeks, followed by a 2-week observation period.
Biological: 1121B — Cohort 6
  13 mg/kg once a week for 4 weeks, followed by a 2-week observation period.
Biological: 1121B — Cohort 7
  16 mg/kg once a week for 4 weeks, followed by a 2-week observation period.

SUMMARY:
The purpose of this study is to determine if IMC-1121B is safe for patients, and to determine the best dose of IMC-1121B to give to patients.

DETAILED DESCRIPTION:
The purpose of this study is to establish the safety profile and the maximum tolerated dose (MTD) of the anti-VEGFR-2 monoclonal antibody IMC-1121B administered weekly in patients with advanced solid tumors who have not responded to standard therapy or for whom no standard therapy is available.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically-documented, measurable or evaluable (non-measurable), advanced primary or recurrent solid tumors who have not responded to standard therapy or for whom no standard therapy is available.
* ECOG performance status score of ≤ 2 at study entry
* Able to provide written informed consent
* A life expectancy of > 3 months
* Adequate hematologic function, as defined by: ANC ≥ 1500/mm^3, hemoglobin level ≥ 10 gm/dL, platelet count ≥ 100,000/mm^3
* Adequate hepatic function, as defined by: total bilirubin level ≤ 1.5 x the ULN, AST and ALT levels ≤ 2.5 x the ULN or ≤ 5 x the ULN if known liver metastases
* Adequate renal function, as defined by a serum creatinine level ≤ 1.5 x the ULN
* Use of effective contraception (per the institutional standard), if procreative potential exists
* Adequate recovery from recent surgery, chemotherapy, and radiation therapy. At least 28 days must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or device, or prior radiation therapy (palliative radiation therapy is allowed).
* Accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center.

Exclusion Criteria:

* Patients with large centrally-located pulmonary lesions adjacent to or invading large blood vessels.
* Patients who have had chemotherapy or therapeutic radiotherapy within 28 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or patients with ongoing side effects ≥ grade 2 due to agents administered more than 28 days earlier.
* Prior left chest wall radiotherapy or a cumulative anthracycline dose ≥ 300mg/m2 (if the ejection fraction is within normal institutional limits, the patient can be enrolled).
* Any concurrent malignancy other than non-melanomatous skin cancer or carcinoma in situ of the cervix. Patients with a previous malignancy but without evidence of disease ≥ 3 years will be allowed to enter the trial.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure, unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months, uncontrolled hypertension, clinically significant cardiac arrhythmia, uncontrolled diabetes, psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements, patients with symptomatic brain metastases
* A serious or nonhealing active wound, ulcer, or bone fracture
* Known HIV positivity
* A major surgical procedure, an open biopsy, or a significant injury within 28 days prior to treatment
* Current or recent use (within 28 days) of a thrombolytic agent
* Current or recent use (within 28 days) of full-dose warfarin
* Chronic daily treatment with aspirin (>325 mg/day) or nonsteroidal anti-inflammatory medications known to inhibit platelet function
* History or clinical evidence of a deep venous or arterial thrombosis (including pulmonary embolism) within 6 months prior to study entry
* Proteinuria ≥1+ by routine urinalysis (patients with a protein value of ≤ 500mg confirmed by a 24-hour urine collection are eligible)
* Pregnant (confirmed by serum beta human chorionic gonadotropin [βHCG]) or breast feeding
* Prior treatment with bevacizumab or other agents specifically targeting VEGF ligand or receptor within 6 weeks of study entry
* Monoclonal antibodies within 6 weeks of study entry
* Positive anti-IMC-1121B antibody response
* History of allergic reactions to monoclonal antibodies or other therapeutic proteins
* Employees of the investigator or study center with direct involvement in this study or other studies under the direction of the investigator or study center, as well as family members the employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | 6 weeks
Maximum Tolerated Dose | 6 weeks

SECONDARY OUTCOMES:
Maximum concentration (Cmax), cohorts 1, 2, 3, 4, 5, 6. and 7 | 6 weeks
Minimum concentration (Cmin), cohorts 1, 2, 3, 4, 5, 6. and 7 | 6 weeks
Area under concentration (AUC), cohorts 1, 2, 3, 4, 5, 6. and 7 | 6 weeks
Half-life (t 1/2), cohorts 1, 2, 3, 4, 5, 6. and 7 | 6 weeks
Clearance (Cl) rate drug is completely removed, cohorts 1, 2, 3, 4, 5, 6. and 7 | 6 weeks
Volume of distribution (Vss) at steady state, cohorts 1, 2, 3, 4, 5, 6. and 7 | 6 weeks
Serum Anti-IMC-1121B Antibody Assessment (immunogenicity) | 6 weeks
Change in tumor size from Baseline Measurement | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (2):
- United States (2):
  - ImClone Investigational Site, Aurora, Colorado
  - ImClone Investigational Site, Philadelphia, Pennsylvania